CLINICAL TRIAL: NCT01813214
Title: Analysis of the Kinetics and Effects of Vemurafenib + Cobimetinib on Intratumoral and Host Immunity in Patients With Advanced BRAFV600 Mutant Melanoma: Implications for Combination With Immunotherapy
Brief Title: The Effects of Vemurafenib + Cobimetinib on Immunity in Patients With Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties.
Sponsor: Georgetown University (Other)
Collaborators: Genentech, Inc. (Industry); Melanoma Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLN28305
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-03

CONDITIONS: Melanoma
Keywords: melanoma; vemurafenib; cobitmetinib
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vemurafenib Monotherapy (Experimental): Vemurafenib 960 mg po BID until unacceptable toxicity or progression of disease
  Interventions: Drug: Vemurafenib
- Vemurafenib + Cobimetinib Combination Therapy (Experimental): Vemurafenib 960 mg po BID until unacceptable toxicity or progression of disease
  Cobimetinib will be given 60mg QD for 21 days on, then 7 days off, in a 28-day treatment cycle.
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: Vemurafenib
  Other Names: Zelboraf; R05185426 (PLX4032)
Drug: Cobimetinib
  Other Names: RO5514041
  Arms: Vemurafenib + Cobimetinib Combination Therapy

SUMMARY:
This study is for patients with malignant melanoma which has spread beyond the local area and cannot be surgically removed, and who have melanoma tumors that are accessible for repeat biopsies. This research study is a way of gaining new knowledge about treatment options for metastatic melanoma. This research study is evaluating the effects of the drugs vemurafenib and cobimetinib on the immune system.

Vemurafenib has been approved by the FDA for treatment of patients with advanced melanoma that harbors a B-RAF mutation. Vemurafenib works by blocking a protein called B-RAF. Researchers have found that a large number of melanomas have mutations (changes) in the BRAF gene. Genes are specific parts of your DNA that contain information on hereditary characteristics such as hair color and eye color. The BRAF gene codes for a protein called B-RAF, which is involved in sending signals in cells that can lead to cell growth. Research has determined that mutations in the BRAF gene at the V600 position cause a change in the B-RAF protein that can drive the growth and spread of melanoma cells.

Cobimetinib (GDC-0973, XL518) is a potent and highly selective inhibitor of MEK1 and MEK2, central components of the RAS/RAF pathway.

The purpose of this research study is to determine how vemurafenib and cobitmetinib may alter the immune system's reaction to melanoma, in order to learn how best to combine immune therapies with vemurafenib in the future.

DETAILED DESCRIPTION:
This is multicenter study of vemurafenib and cobimetinib in patients with biopsy-accessible advanced metastatic melanoma.

The trial will consist of a screening period, a treatment phase, and one post-study follow-up visit occurring about 30 days after the last dose of drug. Day 1 of the study will be defined as the first day a subject receives vemurafenib and/or cobitmetinib. During the treatment phase, all study assessments will be conducted on Day 1 (± 3 days) of each cycle, with the exception of computed tomography (CT) and/or magnetic resonance imaging (MRI), which should occur every 6 weeks (+/- 7 days).

All subjects will have biopsies performed of safely accessible tumors before starting treatment and at 1, 2, and 4 weeks later (days 8, 15, 29). In addition, any patient with accessible tumor at the time of progression will have a tumor biopsy performed at that time.

Mixed-effects models will be used to study the change in CD8 T cell counts per mm^2 of tissue, changes in expression of immunoinhibitory proteins (B7-H1/PD-L1, IDO, arginase), and changes in endothelial homing receptor ligands and tumor associated chemokines at pre-treatment at pre-treatment and at weeks 1, 2, and 4 after therapy. Subjects will be treated as random effects to account for individual variability. Potential covariates are age, gender, and ECOG performance status.

60 ml of blood for lymphocytes will be drawn on days 1, 8, 15, and 29.

ELIGIBILITY:
* Patients must have histological or cytological confirmed melanoma that is metastatic or that is unresectable stage III and clearly progressive.
* Melanoma must be documented to contain a BRAFV600 mutation by a FDA approved assay
* Age > 18 years
* ECOG PS 0,1, or 2
* Participants must have measurable melanoma. Measurable disease is defined as at least one lesion that can be measured accurately in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan. Cutaneous or subcutaneous lesions may be considered measurable if they can be measured reliably as ≥ 10 mm by direct physical exam measurement.

In addition, participants must also have separate disease, which may or may not be measurable as defined by RECIST, but must be readily accessible for core needle biopsy, excisional biopsy, and/or surgical resection. This disease may include one large tumor tissue deposit from which biopsies can be harvested multiple times or may include multiple deposits which can be biopsied, or excised individually, on different dates. Please see below for suggested minimum size requirements of tumor tissue to be used for biopsy for research:

* 1 lesion ≥ 5 cm3 or
* 2 lesions ≥ 3 cm3 each
* 3 lesions ≥ 2 cm3each OR
* ≥ 3 skin lesions, such that the surface area is approximately 1 cm^2 each (or in aggregate for several lesions) and the total volume of tumor I s approximately 260-325 mm^3 or greater for each biopsy time point. These subjects will need ≥ 3 such epidermal/dermal tumor lesions; excisional tumor tissue biopsies will be performed on one or more lesions at each time point. It is acceptable to biopsy more than one lesion, that may be less than 1 cm^2 in surface area, as long as the total tissue removed has a surface area of approximately 1 cm^2 or greater.
* A combination of these may be acceptable, as long as there appears to be enough tumor tissue to remove approximately 325 mm^3 or more of tissue at each time point.

Lesion volume can be calculated based on the formula for volume of a sphere (4/3 r3). An acceptable approximation for lesions approaching spherical shape is to multiply the diameters in three perpendicular directions and divide by 2. [Volume ~ ½(D1xD2xD3); e.g.: volume of a 2 x 2 x 3 cm lesion is approximately 6 cm3. Lesion measurements are based on length X width X depth (height) of sample.]

* Women must not be pregnant due to the fact that the effects of vemurafenib and/or cobimetinib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 6 months after completion of study treatment. See Appendix H for acceptable and unacceptable forms of contraception. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately.
* All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vemurafenib and/or cobimetinib, breastfeeding must be discontinued prior to treatment Day 1 of the study.
* Patients must have measurable disease as defined in Section 9.1. Cutaneous lesions or lymph nodes measuring at least 1 cm will be considered measurable. Baseline CT or MRI scans of measurable disease sites must be performed within 4 weeks of study entry.
* Patients may have received any number of prior systemic treatment regimens for distant metastatic disease or advanced regional disease. The following prior therapy is permitted in either the adjuvant or metastatic disease setting:

  1. No prior therapy
  2. Immunotherapy consisting of interferon-alpha, interleukin-2, GM-CSF, ipilimumab, anti-PD1, cancer vaccines, or other experimental agent.
  3. Cytotoxic chemotherapy consisting of dacarbazine, temozolomide, carboplatin, or paclitaxel alone or in combination.
  4. Targeted therapy with temsirolimus, bevacizumab, or sorafenib.
* Patients who have had prior therapy with a MEK inhibitor or an inhibitor of mutant BRAF are ineligible. Because sorafenib has low efficacy as a BRAF inhibitor, prior therapy with it is allowed.
* Patients must have discontinued cytotoxic therapy agents at least 4 weeks and cytokine and immunoregulatory antibody based immunotherapy at least 6 weeks prior to entering the study and have recovered from adverse events due to those agents.
* Patients must be completed radiation therapy at least 4 week previously
* Patients must have an ECOG performance status of 0, 1 or 2.
* Patients must have the following baseline laboratory values:

  1. White Blood Count > 3,000/mm3
  2. Absolute Granulocyte Count > 1,500/mm3
  3. Platelet Count > 100,000/mm3
  4. Hemoglobin > 9 g/dL
  5. Serum creatinine < 1.5 x upper limit of normal (ULN) or serum creatinine clearance (CrCl) > 40ml/min (CrCl= Wt (kg) x (140-age)*/72 x Cr. level, *female x 0.85)
  6. AST and ALT < 3 x ULN (< 5 x ULN for patients with documented liver metastases)
  7. Alkaline Phosphatase ≤ 2 x ULN (≤ 5x ULN for patients with known liver involvement and ≤ 7x ULN for patients with known bone involvement)
  8. INR < 1.5 and aPTT within 1.1 x ULN. Patients on warfarin therapy are not eligible due to the requirement for multiple biopsies.
  9. Total Bilirubin < 1.5 x ULN
* Patients must not receive any other investigational agents during the period on study or the four weeks prior to entry.
* Patients will be evaluated with a head CT or MRI within 4 weeks of enrollment. Patients must have no clinical evidence of active brain metastasis. Patients with a history of brain metastases must have had them treated greater than 4 weeks previously with the CNS lesions confirmed to be stable or regressing on imaging since the time of the last CNS treatment. Patients must have no residual neurologic symptoms while taking either no steroids or a stable dose of steroids for the 2 weeks prior to enrollment. Patients are allowed to be on a stable dose of anti-seizure meds.
* Patients who have had brain metastases will be eligible only if all of the following are true:

  * the total number of brain metastases ever is ≤ 3
  * all are less than or equal to 2 cm
  * they have been resected surgically or have been treated with gamma-knife or stereotactic radiosurgery
  * the patient has not taken any steroids or has not increased the dose of steroids ≤ 14 days prior to registration.
* Patients must not have another cancer diagnosis with a few exceptions- the following diagnoses will be allowed:

  1. squamous cell cancer of the skin without known metastasis. Note, patients with suspected cuSCCs should have them excised prior to study registration.
  2. basal cell cancer of the skin without known metastasis
  3. carcinoma in situ of the breast (DCIS or LCIS)
  4. carcinoma in situ of the cervix
  5. any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 3 years
* Patients must not have a serious intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring parental antibiotics on Day 1
  * History of congenital long QT syndrome or mean corrected QTc interval > 450 msec at baseline
  * Clinically significant cardiovascular disease:

Myocardial infarction within 6 months Unstable angina New York Heart Association grade II or greater congestive heart failure (see Appendix E) Serious cardiac arrhythmia requiring medication Uncontrolled hypertension ≥ Grade 2 (patients with a history of hypertension controlled with anti-hypertensives to ≤ Grade 1 are eligible) Left ventricular ejection fraction (LVEF) below institutional lower limit of normal or below 50%

* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Psychiatric illness/social situations that would limit compliance with study requirements.

  * Participants must not be known to be HIV positive (testing is not required)
  * Participants must be Hepatitis C negative < 6 months prior to screening
  * Participants must not have a history of malabsorption or other condition that would interfere with absorption of vemurafenib or cobimetinib
  * Patients must be able to comply with study and follow-up procedures.
  * Patients must not have following foods/supplements at least 7 days prior to initiation of and during study treatment: St. John's wort or hyperforin (potent cytochrome P450 CYP34A enzyme inducer) or Grapefruit juice (potent cytochrome P450 CYP34A enzyme inhibitor).
  * Patients must not have significant ocular issues including history of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment, RVO, or neovascular macular degeneration.

The risk factors for RVO are listed below. Patients should be excluded if they have the following conditions:

1. Uncontrolled glaucoma with intra-ocular pressures > 21mmHg
2. Serum cholesterol ≥ Grade 2
3. Hypertriglyceridemia ≥ Grade 2
4. Hyperglycemia (fasting) ≥ Grade 2

   * Patients must have the ability to understand and the willingness to sign a written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Atkins, MD, Principal Investigator — Georgetown Lombardi Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Georgetown Lombardi Comprehsnive Cancer Center, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib Monotherapy: Vemurafenib 960 mg po BID until unacceptable toxicity or progression of disease
  Vemurafenib
- Vemurafenib + Cobimetinib Combination Therapy: Vemurafenib 960 mg po BID until unacceptable toxicity or progression of disease
  Cobimetinib will be given 60mg QD for 21 days on, then 7 days off, in a 28-day treatment cycle.
  Vemurafenib
  Cobimetinib
Period: Overall Study
Arm/Group | Vemurafenib Monotherapy | Vemurafenib + Cobimetinib Combination Therapy
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vemurafenib Monotherapy | Vemurafenib + Cobimetinib Combination Therapy | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time Course by Which Vemurafenib and Cobimetinib Increases T Cell Infiltration
Description: CD8 T cell count per mm^2 of tumor
Time Frame: Day 1, Day 8, Day 15, Day 29
Measure: Mean (Standard Deviation); unit: CD8 T cell count per mm^2 of tumor
Arm/Group | Vemurafenib Monotherapy | Vemurafenib + Cobimetinib Combination Therapy
Number analyzed (Participants) | 3 | 2
CD8 T cell count per mm^2 of tumor
  Day 1 | 7.24 (3.68) | 18.95 (2.64)
  Day 8 | 133.29 (82.22) | 195.77 (185.88)
  Day 15 | 275.08 (125.96) | 51.85 (30.09)
  Day 29 | 197.20 (266.37) | 152.72 (65.54)

2. Primary Outcome: Time Course by Which Vemurafenib and Cobimetinib Increases T Cell Infiltration
Description: CD4 T cell count per mm^2 of tumor
Time Frame: Day 1, Day 8, Day 15, Day 29
Measure: Mean (Standard Deviation); unit: CD4 T cell count per mm^2 of tumor
Arm/Group | Vemurafenib Monotherapy | Vemurafenib + Cobimetinib Combination Therapy
Number analyzed (Participants) | 3 | 2
CD4 T cell count per mm^2 of tumor
  Day 1 | 14.06 (30.36) | 99.12 (18.73)
  Day 8 | 62.17 (40.77) | 51.70 (12.12)
  Day 15 | 186.10 (80.53) | 144.50 (46.65)
  Day 29 | 218.44 (268.82) | 580.1 (419.53)

3. Secondary Outcome: Number of Participants With Tumor Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT and/or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vemurafenib Monotherapy | Vemurafenib + Cobimetinib Combination Therapy
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

ADVERSE EVENTS:
Arm/Group | Vemurafenib Monotherapy | Vemurafenib + Cobimetinib Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vemurafenib Monotherapy (N=3) | Vemurafenib + Cobimetinib Combination Therapy (N=2)
Dehydration (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hyperuricemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Nausea (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Extremity Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Photosensitivity (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Rash-maculopapular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sub-retinal edema (Eye disorders) | 1 (1) | 0 (0)
Elevated ALT (Hepatobiliary disorders) | 1 (1) | 1 (1)
Elevated AST (Hepatobiliary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes